CLINICAL TRIAL: NCT05856058
Title: To Assess SHR0302 Oral Solutions and Tablets in Healthy Subjects Clinical Studies of Relative Bioavailability (Single-center, Random, Open, Crossed)
Brief Title: To Assess SHR0302 Oral Solutions and Tablets in Healthy Subjects Clinical Studies of Relative Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SHR0302-112
Record Dates: First submitted 2023-05-04; First posted 2023-05-12 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Graft-versus-host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — ivarmacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group ARM 1 (Experimental): SHR0302 tablets, then SHR0302 oral solution
  Interventions: Drug: SHR0302
- Treatment group ARM 2 (Experimental): SHR0302 oral solution, then SHR0302 tablets
  Interventions: Drug: SHR0302

INTERVENTIONS:
Drug: SHR0302 — SHR0302 oral solution 1 time, SHR0302 tablets 1 time

SUMMARY:
To assess the relative bioavailability of SHR0302 oral solution and tablet in healthy subjects.

To assess the safety and tolerability of a single dose of SHR0302 oral solution and tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before the start of the activities related to the trial, and be able to understand the procedures and methods of the trial, and be willing to strictly abide by the clinical trial protocol to complete the trial;
2. Age 18~45 years old (including both end values, subject to the signing of informed consent), healthy male;
3. Weight ≥ 50 kg, and body mass index (BMI): 19~26 kg/m2 (including both end values);
4. Sign the informed consent form and agree to use non-pharmacological effective contraception within 60 days after the last dose of the test drug.

Exclusion Criteria:

1. Those who have a history of tobacco addiction within 3 months before signing the informed consent form (an average of 5 cigarettes smoked > per day), or those who cannot stop using any tobacco products during the study;
2. Those who consumed an average of more than 25 g of alcohol per day (e.g., 750 mL of beer, 250 mL of wine, or 50 mL of liquor) per day in the 3 months prior to signing the informed consent form, or who could not stop using any alcohol-containing products during the study, or who had a positive alcohol breath test at screening;
3. Eating any drink or food containing grapefruit within 7 days before randomization; or eat any beverage or food containing methylxanthines, such as coffee, tea, cola, chocolate, etc., within 2 days before randomization;
4. Allergic constitution, or suspected allergy to any ingredient in SHR0302 drug;
5. Drug abusers, or positive urine drug abuse screening at screening, including: morphine, meth (methamphetamine), ketamine, cocaine, ecstasy (MDMA - Methylenedioxymethamphetamine), marijuana (tetrahydrocannabinol acid);
6. Have any history of clinically serious diseases or diseases or conditions that the investigator believes may affect the test results, including but not limited to circulatory, endocrine, nervous system, digestive system, urinary system or blood, immune, psychiatric and metabolic diseases;
7. Those who have a history of tuberculosis within 6 months before signing the informed consent form; or those with a positive γ-interferon release test (IGRA) within 4 weeks prior to randomization;
8. 12-lead ECG QTcF > 450 ms or other abnormalities judged clinically significant by the investigator in the first 4 weeks of randomization;
9. Vital signs, physical examination, laboratory tests, abdominal ultrasound or chest imaging in the first 4 weeks of randomization suggest that there are abnormalities that are judged to be clinically significant by the investigator;
10. Within 4 weeks before randomization, hepatitis B surface antigen (HBsAg) positive, or anti-hepatitis C virus (HCV) antibody positive, or human immunodeficiency virus (HIV) antibody positive, or syphilis antibody positive;
11. Infections (viral, bacterial, fungal, parasitic infections) that require systemic antimicrobial therapy within 4 weeks of randomization;
12. Use of any prescription drug, over-the-counter drug, Chinese herbal medicine or dietary supplement within 2 weeks prior to randomization;
13. Systemic therapy with inhibitors or inducers of cytochrome P450 3A4 enzyme (CYP3A4) within 4 weeks before randomization (see Annex 2 for details);
14. Those who participated in any drug clinical trial and took the experimental drug within 3 months before randomization (calculated from the start time of the last visit of the last trial) (if the 5 half-lives of the experimental drug exceed 3 months, the time of the 5 half-lives shall prevail);
15. Have received BCG vaccine within 12 months prior to randomization; or vaccination or exposure to other live vaccines or live attenuated vaccines within the first 3 months of randomization; or those who plan to be vaccinated during the trial;
16. Those who have undergone any surgery within the previous 3 months of randomization, or who have not recovered after surgery, or who may have surgery or hospitalization plans during the estimated trial period;
17. Those who donate blood (or lose blood) within 3 months of randomization and donate blood (or blood loss) in an amount ≥ 400 mL, or receive blood transfusion;
18. The investigator judges that the subject has a situation that affects the absorption, distribution, metabolism and excretion of drugs, or has other factors that are not suitable to participate in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
SHR0302 and its main Pk parameter, AUC0-t | day 1 to 8
SHR0302 and its main Pk parameter, AUC0-inf | day 1 to 8
SHR0302 and its main Pk parameter, Cmax | day 1 to 8
Relative bioavailability (F%) value between SHR0302 oral solution and SHR0302 tablet: F% = AUC0-t (oral solution) / AUC0-t (tablet) ×100% | day 1 to 8

SECONDARY OUTCOMES:
SHR0302 and its main Pk parameter, Tmax (SHR0302 only) | day 1 to 8
SHR0302 and its main Pk parameter, t1/2 (SHR0302 only) | day 1 to 8
SHR0302 and its main Pk parameter, CL/F (SHR0302 only) | day 1 to 8
SHR0302 and its main Pk parameter, Vz/F (SHR0302 only) | day 1 to 8
Adverse events | day 1 to 12

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided